CLINICAL TRIAL: NCT05784259
Title: Development and Clinical Trial of a Transdiagnostic Single-session Treatment for Primary Care Patients
Brief Title: Development of Transdiagnostic Single-session Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luleå Tekniska Universitet (Other)
Collaborators: Region Norrbotten (Unknown)
Responsible Party: Principal Investigator, John Näsling, Lic. psychologist / Doctoral student, Luleå Tekniska Universitet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 275863
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Anxiety Disorders; Depression; Stress Disorder
Keywords: transdiagnostic; single-session
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- Treatment group (Experimental): Transdiagnostic single-session treatment
  Interventions: Behavioral: Transdiagnostic single-session treatment

INTERVENTIONS:
Behavioral: Transdiagnostic single-session treatment — Administered over 4 hour in group of 10 patients. Interventions are: Psychoeducation of emotions, De-fusion exercise, Mindfulness exercise, Interoceptive exposure, Behavioral activation
  Arms: Treatment group

SUMMARY:
The goal of this clinical trial is to test a single session treatment program in primary care patients with anxiety and/or depression and/or stress-related issues. The main questions it aims to answer is:

* Will the transdiagnostic treatment program decrease symptoms of depression/anxiety/stress?
* Will the transdiagnostic treatment program decrease transdiagnostic risk factors?
* Will the transdiagnostic treatment program decrease the measured risk factors equally?
* Will the transdiagnostic treatment program impact patients with anxiety, depression or stress disorders equally?
* Will the transdiagnostic treatment program have long term (6 months post-treatment) effect on transdiagnostic risk factors?
* Will the transdiagnostic treatment program have long term (6 months post-treatment) effect on anxiety, depression, or stress-symptoms?
* Have the participants been able to generalize the skills taught in the program(qualitative)?
* Within group that were treated with single-session treatment and recieved additional care before follow-up, was there a difference in outcome?

DETAILED DESCRIPTION:
The study investigates the effect of a single-session, 4 hour, transdiagnostic treatment for primary care patientst with depression, anxiety or stress.

The treatment includes, interoceptive exposure, behavioral activation, mindfulness, defusion and psycho-education about emotions.

The study is conducted in a clinical setting in northern sweden and follows up results at 3 weeks and 6 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for anxiety, mood disorder, or stress diagnosis
* Symptoms are mild to moderate in severity

Exclusion Criteria:

* Already in ongoing psychotherapy
* Within a month commenced pharmaceutical treatment that will likely impact mood or psychological functioning and is not deemed to be on a stable dose
* Has a comorbid personality disorder
* Has a risk of suicide deemed other than low
* Has other severe psychological disorders outside the scope of primary care
* Is in a severely stressful social situation deemed incompatible with psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety, Depression and Stress symptoms post-treatment | 3 weeks post-treatment
  Measured using DASS-21
Anxiety, Depression and Stress symptoms follow-up | 6 months post-treatment
  Measured using DASS-21
Anxiety sensitivity post-treatment | 3 weeks post-treatment
  Measured using BSQ, fear of bodily sensations related to anxiety
Anxiety sensitivity follow-up | 6 months post-treatment
  Measured using BSQ, fear of bodily sensations related to anxiety
Experiential avoidance post-treatment | 3 weeks post-treatment
  Measured using AFQ-Y8, psychological flexibility
Experiential avoidance follow-up | 6 months post-treatment
  Measured using AFQ-Y8, psychological flexibility
Mindfulness post-treatment | 3 weeks post-treatment
  Measured using FFMQ, mindfulness
Mindfulness follow-up | 6 months post-treatment
  Measured using FFMQ, mindfulness
Alexithymia post-treatment | 3 weeks post-treatment
  Measured using TAS-20, mindfulness
Alexithymia follow-up | 6 months post-treatment
  Measured using TAS-20, mindfulness
Generalization | 6 months post-treatment
  Qualitative interview with a few selected patients to review their experience of the treatment, its effectiveness and their ability to use the techniques taught.

SECONDARY OUTCOMES:
Additional treatment | 6 months post-treatment
  It will be recorded if patients sought additional care after single-session treatment as well as type of care.

CONTACTS AND LOCATIONS:
Overall Officials: John Näsling, Master, Principal Investigator — Luleå tekniska universitet/Region Norrbotten
Locations (1):
- Region Norrbotten, Primary care, Luleå, Norrbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No